CLINICAL TRIAL: NCT07341659
Title: A Multicentric, Randomized, Blinded, Comparative Study to Evaluate the Efficacy of the Cosmetic Product RV3278B-OS0386 in the Maintenance Phase After Oral Isotretinoin Treatment of Adult Subjects With Facial Acne.
Brief Title: Efficacy of Cosmetic Product RV3278B-OS0386 in the Maintenance Phase After Oral Isotretinoin Treatment of Adults Subjects With Facial Acne.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RV3278B20240495
Record Dates: First submitted 2025-12-15; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Acne
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): This group will apply the test cosmetic product
  Interventions: Other: Test product RV3278BB-OS0386
- Control Group (Placebo Comparator): This group will apply the control cosmetic product
  Interventions: Other: Control product RV3278B-OS0548

INTERVENTIONS:
Other: Test product RV3278BB-OS0386 — Cosmetic product RV3278BB-OS0386 to be applied twice a day on the face during the whole study
  Arms: Test Group
Other: Control product RV3278B-OS0548 — Cosmetic product RV3278B-OS0548 to be applied twice a day on the face during the whole study
  Arms: Control Group

SUMMARY:
The aim of this study is to evaluate the efficacy of the RV3278B-OS0386 cosmetic product, compared to the control product in managing acne relapse during the 12-month maintenance phase follow-up after oral isotretinoin treatment in adult subjects with facial acne.

DETAILED DESCRIPTION:
This study is conducted as a multicentric, randomized, blinded, comparative study in Europe.

A total number of 102 subjects included and randomized in 2 parallel groups:

* Test group: twice daily application of the RV3278B-OS0386 cosmetic product on the whole face
* Control group: twice daily application of the RV3278B-OS0548 cosmetic product on the whole face

Subjects will be followed at regular intervals for up to 12 months or until the relapse of their acne on the face, whichever occurs first.

6 visits are planned:

* Visit 1 (Day 1): Inclusion, Randomization and start of product
* Visit 2 (month 1)
* Visit 3 (month 3)
* Visit 4 (month 6)
* Visit 5 (month 9)
* Visit 6 (month 12): End of study Visit In case of subject's acne relapse confirmed by the investigator, subject will be withdrawn from the study.

As part of an ancillary exploratory assessment, outcome measures will also be evaluated on augmented datasets including both study subject's data and synthetic data generated from the study subject's data by artificial intelligence.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged between 15 and 35 years included
* Subject affiliated to a social security system or health insurance, or is a beneficiary if applicable
* Subject who recently completed his/her first course of oral isotretinoin treatment
* Subject with clear or almost clear facial acne

Non Inclusion criteria:

* Subject who, in the judgement of the investigator, is not likely to be compliant with study-related constraints and requirements
* Facial skin disease other than acne, skin abnormalities, or dermatological condition on the face liable to interfere with the study assessments
* Severe or complicated cases of acne (ex: acne conglobate) according to investigator's assessment
* Any acute, chronic or progressive disease or medical history liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
* Any surgery, chemical (e.g.: skin peel) or physical treatment on the face done within 12 months before the inclusion or planned during the study
* Topical or systemic product or treatment established or modified during the previous weeks or planned to be established or modified during the study, liable to interfere with the evaluation of the efficacy or cutaneous tolerance of the investigational product according to the investigator's assessment

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Actual)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Acne relapse rate | From Visit 1 (Day 1) to Visit 6 (Month 12 or early termination )
  The acne relapse rate is defined as percentage of subjects experiencing acne relapse on the face according to the investigator

SECONDARY OUTCOMES:
Acne severity by investigator | Visit 1 (Day 1),Visit 2 (Month 1), Visit 3 (Month 3), Visit 4 (Month 6), Visit 5 (Month 9) and Visit 6 (Month 12 or early termination).
  Acne severity will be assessed by the investigator on the face using a 6-point scale (0 to 5 with 0: clear and 5: very severe)
Time to acne relapse | From Visit 1 (Day 1) to Visit 6 (Month 12 or early termination)
  Time to acne relapse will be calculated from the date of the visit 1 until the date of the acne relapse as assessed by the investigator.
Acne lesions count | Visit 1 (Day 1), Visit 2 (Month 1), Visit 3 (Month 3), Visit 4 (Month 6), Visit 5 (Month 9) and Visit 6 (Month 12 or early termination).
  Assessed by the investigator according to the Lucky Method by counting papules, pustules, open and closed comedones on the face
Post-inflammatory lesions count | Visit 1 (Day 1), Visit 2 (Month 1), Visit 3 (Month 3), Visit 4 (Month 6), Visit 5 (Month 9) and Visit 6 (Month 12 or early termination).
  Assessed by the investigator by counting post-inflammatory hyperpigmentation and erythema lesions on the face
Acne severity by subject | Visit 1 (Day 1), Visit 2 (Month 1), Visit 3 (Month 3), Visit 4 (Month 6), Visit 5 (Month 9) and Visit 6 (Month 12 or early termination), and monthly at home.
  Acne severity will be assessed by the subject on the face using a 7-point scale (-3 to 3 with -3: much worse and 3: much improved)
Quality of life questionnaire | Visit 1 (Day 1), Visit 3 (Month 3) and Visit 6 (Month 12 or early termination).
  Quality of life will be assessed by the subject by completing the Cardiff Acne Disability Index Questionnaire consisting in 5 questions, each response is on a 4-point scale.
Adverse events | From Visit 1 (Day 1) to Visit 6 ( Month 12 or early termination)
  Adverse events occurrence will be determined by the subject or subject's/parent(s) or guardian(s) spontaneous reporting, the investigator's non-leading questioning and his/her clinical evaluation
Global Tolerance | Visit 3 (Month 3) and Visit 6 (Month 12 or early termination).
  Global Tolerance will be assessed by the investigator with 5-point scale (from 0: bad to 5: excellent)
Acceptability Questionnaire assessment | Visit 4 (Month 6) and Visit 6 (Month 12 or early termination).
  Acceptability questionnaire regarding the use of the product will be completed by the subject.
Standardized photographs of the subject's face for illustrative purpose only | Visit 1 (Day 1), Visit 4 (Month 6), and Visit 6 (Month 12 or early termination).
  for illustrative purpose only
Transepidermal water loss | Visit 1 (Day 1), Visit 2 (Month 1), Visit 3 (Month 3), Visit 4 (Month 6), Visit 5 (Month 9) and Visit 6 (Month 12 or early termination).
  Transepidermal water loss measurement by Tewameter.
Skin potential hydrogen | Visit 1 (Day 1), Visit 2 (Month 1), Visit 3 (Month 3), Visit 4 (Month 6), Visit 5 (Month 9) and Visit 6 (Month 12 or early termination).
  Skin potential hydrogen measurement by pH meter.

CONTACTS AND LOCATIONS:
Locations (5):
- Centre de santé Sabouraud, Paris, France
- Italy (2):
  - Humanitas Research Hospital - Unita dermatologica, Milan
  - Istituto Dermopatico dell'Immacolata in Roma, Roma
- Poland (2):
  - Dr. E.Karamon Private Practice, Malbork, Poland
  - Dr. I.Karamon Private Practice, Gdansk